CLINICAL TRIAL: NCT06374875
Title: A Prospective Multicenter International Randomized Controlled Trial Comparing Surgical and Medical Therapies in the Treatment of Advanced Metabolic Dysfunction Associated Steatohepatitis
Brief Title: Fibrosis Lessens After Metabolic Surgery
Acronym: FLAMES
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ali Aminian (Other)
Collaborators: Sobia Laique, MD (Unknown)
Responsible Party: Sponsor-Investigator, Ali Aminian, Director of Bariatric and Metabolic Institute, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-213
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD); Non-Alcoholic Fatty Liver Disease; Metabolic Dysfunction-Associated Steatohepatitis (MASH); Liver Fibrosis; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Obesity | interventions — Bariatric Surgery; Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio into 1 of the 2 arms using a computer-generated randomization plan, stratified to ensure that there are equal number of patients with/without T2DM and with/without F4 (cirrhosis) according to the baseline liver biopsy in each treatment group (surgical group vs non-surgical group). The participant sites are regrouped into three geographic regions. All patients in each region will be randomized separately to have equal number of patients with/without T2DM and with/without F4 in each treatment group in each region.
Who Masked: Outcomes Assessor
Masking Description: Patients and investigators will not be blinded to treatment assignment. The treatment assignment will remain unknown until the patient is randomized after meeting all eligibility requirements.
  Pathologists who report the liver biopsies (to assess the primary end point of study) are blinded to treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metabolic Surgery (Active Comparator): FLAMES will examine the class effect (not the specific procedure effect) of metabolic surgery. The study is not intended to compare Roux-en-Y Gastric Bypass (RYGB) vs Sleeve Gastrectomy (SG) head-to-head. RYGB and SG constitute one group as a metabolic surgery group. Assignment of RYGB or SG is not based on a randomized design. Each patient and surgical team will make a shared decision about the most appropriate surgical procedure.
  Interventions: Procedure: Metabolic surgery
- Incretin-Based Therapy (Active Comparator): Three incretin-based medications that have been approved for treatment of obesity including liraglutide, semaglutide, or tirzepatide will be used in the nonsurgical group. The FLAMES will examine the class effect (not the specific drug effect) of incretin-based therapies. The study is not intended to compare semaglutide vs tirzepatide vs liraglutide head-to-head.
  Interventions: Drug: Incretin-Based Therapy

INTERVENTIONS:
Procedure: Metabolic surgery — Patients receive either RYGB or SG. The surgical risk, differential impact of each procedure on body weight and other obesity-related diseases, presence of other medical and mental problems, patient's behavioral factors (e.g., postoperative compliance, active smoking), medications, and goals will be considered when the patient and local medical team make a shared decision about the most appropriate surgical procedure
  Other Names: Bariatric surgery; Roux-en-Y Gastric Bypass (RYGB); Sleeve Gastrectomy (SG)
  Arms: Metabolic Surgery
Drug: Incretin-Based Therapy — Three incretin-based medications that have been approved for treatment of obesity including liraglutide, semaglutide, or tirzepatide will be used in the nonsurgical group. Any of these 3 medications (in the injection or oral from) based on availability in each country, access, and clinical indications can be used. If possible, patients will be placed on high-dose tirzepatide (Mounjaro or Zepbound 15 mg once weekly injection) or high-dose semaglutide (Wegovy 2.4 mg once weekly injection or Ozempic 2 mg once weekly injection). Other acceptable, less preferrable, options: liraglutide (Saxenda or Victoza), semaglutide tablet (Rybelsus), or lower dose of tirzepatide and semaglutide injections.
  Other Names: Glucagon-like Peptide-1 Receptor Agonist
  Arms: Incretin-Based Therapy

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD), formerly known as non-alcoholic fatty liver disease (NAFLD), a major global public health concern, is commonly associated with obesity, diabetes, and dyslipidemia. MASLD is currently the most common cause of chronic liver disease affecting about 80% of people with obesity, ranging from simple fat deposits in the liver to Metabolic Dysfunction-Associated Steatohepatitis (MASH), cellular injury, advanced fibrosis, cirrhosis, or hepatocellular carcinoma. Patients with MASH are also at risk for cardiovascular disease and mortality. There is no universally approved medication for MASH. Weight loss remains the cornerstone of MASH treatment.

Patients meeting the inclusion and exclusion criteria and who give informed consent will be enrolled in the trial and undergo the baseline liver biopsy (if none available). Approximately 120 patients with MASH and liver fibrosis (F1-F4 in baseline liver biopsy) will be randomized in a 1:1 ratio to metabolic surgery or medical treatment (incretin-based therapies ± other medical therapies for MASH) and followed for 2 years at which time a repeat liver biopsy will be performed for the assessment of the primary end point.

DETAILED DESCRIPTION:
FLAMES (Fibrosis Lessens After Metabolic Surgery) is a 2-arm randomized, controlled, pathologist-blinded multicenter study with 2 parallel groups of patients with MASH, liver fibrosis, and obesity who will either receive metabolic surgery or incretin-based therapies (semaglutide [injection or oral], tirzepatide [injection], or liraglutide [injection]) for 2 years to assess the effects of advanced surgical and medical therapies in liver histology in patients with obesity, biopsy-proven MASH, and liver fibrosis. With genuine uncertainty in the expert medical community and literature over which treatment will result in a greater improvement in histopathological features of MASH and liver fibrosis, the investigators aim to compare metabolic surgery and incretin-based therapies head-to-head.

Adult patients with BMI between 35 - 60 kg/m^2, Fibrosis-4 (FIB-4) index ≥ 1.3, liver stiffness measure (LSM) ≥ 12 kPa by vibration-controlled transient elastography (VCTE) using FibroScan (or similar non-invasive tests) who meet the contemporary eligibility criteria for metabolic surgery will be eligible for participation. Patients meeting the inclusion and exclusion criteria and who give informed consent will be enrolled in the trial and undergo the baseline liver biopsy. Approximately 120 patients with MASH and liver fibrosis (F1-F4 in baseline liver biopsy) will be randomized in a 1:1 ratio to metabolic surgery or medical treatment (incretin-based therapies ± other medical therapies for MASH) and followed for 2 years at which time a repeat liver biopsy will be performed for the assessment of the primary end point.

The primary site of this multicenter, international, randomized controlled trial (RCT) is at the Cleveland Clinic main campus in Cleveland, Ohio, USA.

ELIGIBILITY:
Inclusion Criteria

Entry into the study would require that the patient:

1. Is a candidate for general anesthesia
2. Is eligible for metabolic surgery (RYGB or SG) based on the ASMBS/IFSO 2022 guidelines
3. Has insurance coverage for metabolic surgery (the requirements may vary in each country)
4. Is ≥18 and ≤75 years old at the time of signing the informed consent
5. Has a BMI ≥35 and ≤70 kg/m2 at the time of first study visit
6. FIB-4 ≥ 1.3
7. At least one of the following 5 criteria suggesting presence of advanced fibrosis:

   * LSM ≥ 12 kPa by VCTE using FibroScan®
   * LSM ≥ 12 kPa by SWE
   * LSM ≥ 1.7 m/s by ARFI
   * LSM ≥ 3.63 kPa MRE
   * ELF score ≥ 9.8
8. Patients with and without T2DM are eligible for the study. Patients with T2DM should have been on a stable dose of anti-diabetic medication (including insulin but not semaglutide or tirzepatide or liraglutide) for at least 3 months prior to entry, with glycated hemoglobin (HbA1c) ≤12%.
9. Self-reported stable weight in 6 months before the first study visit (no weight loss >10% within 6 months prior to the first study visit)

   a. In patients with a historical noninvasive tests or liver biopsy, weight loss of no more than 10% is allowed from 6 months prior to the historical tests until the first study visit
10. Has the ability and willingness to participate in the study, provide informed consent, and agree to any of the arms involved in the study
11. Can understand the options and comply with the requirements of each arm, including one liver biopsy performed during the screening period (if no adequate biopsy within 12 months before screening is available) and one liver biopsy after 2-years
12. Has a negative urine pregnancy test at the first and at the randomization visits for women of childbearing potential.
13. Women of childbearing age must agree to use reliable method of contraception for 2 years

8.2 Exclusion Criteria

Patients who meet the following criteria will be excluded from the study:

1. Known history of other chronic liver diseases (drug induced, viral hepatitis, autoimmune, and genetic):

   * Hepatitis B as detected by presence of hepatitis B surface antigen (HBsAg)
   * Hepatitis C as detected by presence of hepatitis C virus (HCV) RNA (in case the screening test for hepatitis C is positive, the confirmative test is decisive)
   * Autoimmune liver disease as diagnosed by antibodies or compatible liver histology
   * Primary biliary cirrhosis as defined by the presence of at least 2 criteria (elevated alkaline phosphatase, presence of anti-mitochondrial antibody, and histologic evidence of nonsuppurative destructive cholangitis and destruction of interlobular bile ducts)
   * Primary sclerosing cholangitis
   * Wilson's disease as diagnosed by low ceruloplasmin or compatible liver histology
   * Alpha-1-antitrypsin deficiency as diagnosed by alpha1-antitrypsin level or liver histology
   * Hemochromatosis as diagnosed by HFE mutations (C282Y, H63D), ferritin and transferrin saturation levels, or presence of 3+ or 4+ stainable iron on liver biopsy
   * Drug-induced liver disease diagnosed by medical history
   * Known bile duct obstruction
   * Suspected or proven liver cancer
2. Weight change >10% within 6 months prior to the first study visit or prior to the historical liver biopsy
3. Treatment with semaglutide, tirzepatide, or liraglutide (for obesity or for T2DM) <90 days before the first study visit.

   • However, patients are allowed to participate if they have been on a low dose (or are on older generation GLP-1 agonists) and have lost less than 10% of their body weight since starting the medication.
4. Type 1 diabetes or autoimmune diabetes
5. Known cases of human immunodeficiency virus infection
6. Prior bariatric and metabolic surgery of any kind

   • Reversed procedures such as gastric band or intragastric balloon that have been removed at least 3 months prior to the first study visit are allowed.
7. Prior complex foregut surgery including any esophageal and gastric surgeries, anti-reflux procedures, biliary diversion, and complex trauma surgery
8. Any surgery requiring general anesthesia within 1 month prior to signing the consent
9. History of solid organ transplant
10. Severe pulmonary disease defined as FEV1 < 50% of predicted value
11. Significant cardiac or atherosclerotic disease (planned to undergo cardiac, coronary, carotid, or peripheral artery revascularization procedures in the next 12 months)
12. Severe uncompensated cardiopulmonary disease leading to American Society of Anesthesiologists Class IV or V
13. Classified as New York Heart Association Class IV
14. Left ventricular ejection fraction <25% at the time of screening
15. Myocardial infarction, unstable angina, stroke, heart surgery, coronary stent placement in the past 6 months
16. Chronic renal insufficiency with eGFR below 30 mL/min/1.73 m2, or being on dialysis
17. Presence of large hiatal hernia (>7 cm)
18. Presence of Crohn's disease
19. Psychiatric disorders including (but not limited to) dementia, active psychosis, severe depression requiring 3 or more medications, history of suicide attempts, active alcohol, or substance abuse within the previous 12 months that in the opinion of the investigators could disqualify the patient from metabolic surgery
20. Pregnancy, the intention of becoming pregnant, or not using adequate contraceptive measures
21. Breastfeeding
22. Diagnosis of malignancy within the preceding 3 years (except squamous cell and basal cell cancer of the skin)
23. Anemia defined as hemoglobin less than 9 g/dL
24. On therapeutic dose of anticoagulants such as warfarin or direct oral anticoagulants (DOACs)
25. Known history of clotting disorders, including pulmonary embolus and deep vein thrombosis
26. Clinical judgment that life expectancy is less than 3 years
27. Use of investigational therapy within 3 months prior to signing the consent
28. History of pancreatic carcinoma
29. Acute pancreatitis < 180 days before screening
30. History or presence of chronic pancreatitis
31. Presence of concerning thyroid nodule
32. Uncontrolled thyroid disease: thyroid stimulating hormone (TSH) > 6.0 mIU/L or < 0.1 mIU/L before the first study visit

    * Patients receiving treatment for hypothyroidism can be included if their thyroid hormone replacement dose has been stable for at least 3 months.
    * Patients whose TSH is outside the rang but they have normal levels of thyroid hormones can be included.
33. A personal or family history of medullary thyroid carcinoma (MTC) or in patients with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
34. Evidence or history of ascites or spontaneous bacterial peritonitis that require(d) treatment

    • Trace ascites identified only by an abdominal imaging without other evidence of clinically significant portal hypertension and esophageal varices is not an exclusion criterion.
35. Evidence or history of hepatic encephalopathy
36. Evidence or history of variceal bleeding
37. Evidence or history of portosplenic vein thrombosis
38. Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to the first study visit.

    • Defined as more than 14 units/week for females (>1 drink per day) and more than 21 units/week for males (>2 drinks per day) on average, where one unit of alcohol is equivalent to a 12-oz beer, 4-ounce glass of wine, or 1-ounce shot of hard liquor.
39. Treatment with medications (for more than 14 consecutive days) with known effect on liver steatosis (e.g., treatment with systemic corticosteroids [oral or intravenous], methotrexate, tamoxifen, valproic acid, amiodarone, or tetracycline) in the 3 months prior to the first study visit (or historical liver biopsy).
40. ALT or AST or Alkaline phosphatase >200 U/L
41. Recurrent major hypoglycemia or hypoglycemic unawareness
42. Inability to safely obtain a liver biopsy
43. Any condition or major illness that, in the investigator's judgment, places the subject at undue risk by participating in the study
44. Unable to understand the risks, benefits, and compliance requirements of study
45. Lack capacity to give informed consent
46. Plans to move outside the primary location of study (country) within the next 24 months
47. Known or suspected allergy to semaglutide, tirzepatide, liraglutide, excipients, or related products
48. Previous participation in this trial and got randomized to one of the study groups but did not proceed.
49. Hospitalization due to COVID-19 within 2 months prior to screening.
50. Platelet count <80,000
51. International Normalized Ratio (INR) >1.7
52. Child-Pugh score B or C
53. MELD score ≥15
54. Upper endoscopy showing gastroesophageal varices
55. Upper endoscopy showing more than mild portal hypertensive gastropathy
56. Liver vascular ultrasound (duplex ultrasonography) showing significant portal hypertension characterized by dilated portal vein (>13 mm), biphasic or reverse flow in the portal vein, enlarged paraumbilical veins, splenorenal collaterals, or dilated left and short gastric veins.

    Note: Negative findings on upper endoscopy and liver duplex ultrasound (done within one year of the first study visit for both tests) are necessary to establish eligibility for the FLAMES.
    * Ruling out clinically significant portal hypertension is particularly important in patients with a liver stiffness ≥20 kPa or with a platelet count <150,000 per μL or with a (historical) liver biopsy showing cirrhosis.
    * A subset of patients without having upper endoscopy and liver duplex ultrasound can be eligible for enrollment if their:

      * liver stiffness (by transient elastography using FibroScan®) is between 12 and 15 kPa and their platelet count is >150,000 per μL, or
      * a (historical) liver biopsy showing absence of cirrhosis, or
      * a (historical) HVPG < 5 mmHg
57. Cross-sectional abdominal imaging (if available historically) indicating presence of large portosystemic collaterals or ascites

    • Splenomegaly alone (in the absence of other radiological and laboratory findings) is not considered to be a sign of clinically significant portal hypertension and is not an exclusion criterion.
58. HVPG ≥ 12 mmHg (if available historically or if measured at the time of de novo liver biopsy)
59. Liver biopsy characteristics:

    * F0 in de novo biopsy; Enrollment cap of 20% for F1 in de novo biopsy.
    * F0 and F1 in historical liver biopsy
    * Absence of all three components of MASH (steatosis, hepatocyte ballooning, and lobular inﬂammation) in patients with F1, F2, and F3
    * Absence of steatosis (<5%) in patients with F4
    * Diagnosis other than MASH

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of at least 1 fibrosis stage of the Kleiner fibrosis classification and no worsening of MASH in the repeat liver biopsy. | Through study completion, 2 years
  Development of hepatic decompensation events including ascites (requiring treatment including diuretics), spontaneous bacterial peritonitis, hepatic encephalopathy (requiring treatment or hospitalization), or bleeding esophageal varices, and all-cause mortality will be counted as a treatment failure with no need for repeating liver biopsy.

SECONDARY OUTCOMES:
MASH resolution in the repeat liver biopsy | Through study completion, 2 years
  MASH resolution defined as no hepatocyte ballooning (score of 0 according to the NASH CRN criteria), no more than mild residual inflammatory cells (score of 0 or 1), without worsening of liver fibrosis stage in the repeat liver biopsy
MASH resolution and fibrosis improvement in the repeat liver biopsy | Through study completion, 2 years
  Presence of both MASH resolution and fibrosis improvement in the repeat liver biopsy
Fibrosis progression in the repeat liver biopsy | Through study completion, 2 years
  Defined as worsening of at least 1 fibrosis stage of the Kleiner fibrosis classification in the repeat liver biopsy among patients who did not have F4 in the baseline liver biopsy
Average Weight loss percentage | Through study completion, 2 years
  Mean percentage weight loss from baseline
Disease-specific Quality of Life (QoL) | Through study completion, 2 years
  Change from baseline in score of a disease-specific QoL instrument: Chronic Liver Disease Questionnaire (CLDQ) for NASH (CLDQ-NASH). This instrument collects data on 36 items grouped into 6 domains: abdominal symptoms, activity/energy, emotional health, fatigue, systemic symptoms, and worry. In all domains, greater scores (between 1-7) reflect better health, and the average of the domain scores yields the total CLDQ-NASH score. Research coordinator completes the survey with the patient.

OTHER OUTCOMES:
MASLD-related histopathologic end points | Through study completion, 2 years
  * Improvement of at least 1 fibrosis stage of the Kleiner fibrosis classification, regardless of changes in MASH severity
  * Progression to cirrhosis (F4) in repeat liver biopsy among patients who did not have F4 in the baseline liver biopsy
  * Mean and change from baseline in NAFLD Activity Score
  * Reduction in NAFLD Activity Score by at least 1, 2, or 3 points
  * Histopathological changes in severity of steatosis, inflammation, hepatocyte ballooning, and fibrosis
  * Histopathological changes in modified Ishak fibrosis score
  * Histopathological changes in features of regression (Beijing classification, P-I-R fibrosis quality)
MASLD-related laboratory end points | Through study completion, 2 years
  Mean and change from baseline in ALT, AST, Alkaline phosphatase, bilirubin, platelet count, eGFR, and FIB-4
MASLD-related liver scan end points | Through study completion, 2 years
  Change in liver stiffness in elastography (based on the same device that was used at baseline)
MASLD-related clinical end points | Through study completion, 2 years
  Development of adverse clinical outcomes including development of ascites or hydrothorax (requiring treatment including diuretics), hepatic encephalopathy (requiring treatment or hospitalization), bleeding esophageal varices, liver-related mortality, and all-cause mortality as a composite and individual end points
Achieved Weight-loss proportions | Through study completion, 2 years
  Proportion of participants achieving ≥ 5%, ≥ 10%, ≥ 15%, ≥ 20%, ≥ 25%, ≥ 30%, ≥ 35% weight loss from baseline (yes/no) in each two groups
Weight change (kg) | Through study completion, 2 years
  Absolute change in weight (kg)
BMI change (kg/m^2) | Through study completion, 2 years
  Absolute change in BMI (kg/m^2)
Excess weight loss, % | Through study completion, 2 years
  Calculated by dividing the difference between initial BMI and final BMI by the difference between initial BMI and a target BMI of 25
Change in waist circumference, cm | Through study completion, 2 years
  Change in circumferential measurement above the level of the iliac crests
Systolic blood pressure trends, mmHg | Through study completion, 2 years
  Mean and change in systolic blood pressure, mmHg
Mean and change from baseline in lipid panel, mg/dl | Through study completion, 2 years
  Mean and change from baseline in total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), and triglycerides
Changes in glucose hemostasis markers | Through study completion, 2 years
  Mean and change from baseline in blood glucose, HbA1c, and fasting homoeostasis model of assessment of insulin resistance (HOMA-IR) in patients with T2DM
Percentage of patients with T2DM meeting predefined HbA1c targets | Through study completion, 2 years
  * HbA1c <6.5% (without diabetes medications)
  * HbA1c <7% (irrespective of taking diabetes medications or not)
Changes in inflammatory markers, CRP mg/L | Through study completion, 2 years
  Mean and change from baseline in C-Reactive Protein (CRP)
Change in cardiovascular and diabetes medications | Through study completion, 2 years
  Change in number of cardiovascular and diabetes medications prescribed
SF-Bari Score | Through study completion, 2 years
  Swiss-Finnish Bariatric Metabolic Outcome Score (SF-BARI Score) which combines four areas of clinical interest in obesity treatment (weight loss, outcomes of four major obesity-related comorbidities, complications, and QoL) in one score. The SF-BARI Score range is from -100 to 200 and the SF-BARI Score QOL is from -130 to 230. The total score ranges from suboptimal (scores below 35) to excellent (scores equal or greater than 135). Research coordinator completes the survey with the patient.
Quality of life end points | Through study completion, 2 years
  Change from baseline in score of The 36-Item Short Form Health Survey (SF-36) (physical and mental components). Each item is given a score ranging from 0-100. Lower scores indicating poor outcomes. Final score is an average of all the items that were answered. Unanswered questions are not included in the final average. Research coordinator completes the survey with the patient.
Safety end points | Through study completion, 2 years
  Complications specifically related to MASH disease, as well as complications of liver biopsy, metabolic surgery, liraglutide, semaglutide, tirzepatide, and other medications will be recorded and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Aminian, MD, Principal Investigator — The Cleveland Clinic
Locations (22):
- United States (4):
  - Banner Health Center, Phoenix, Arizona
  - Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
- Hospital Alemão Oswaldo Cruz, São Paulo, Brazil
- McGill University, Montreal, Canada
- Turku University Hospital, Turku, Finland
- India (2):
  - Sri Aurobindo Institute of Medical Sciences, Indore
  - The Digestive Health Institute, Mumbai
- University College Dublin, Dublin, Ireland
- Italy (2):
  - Università Cattolica del Sacro Cuore, Milan
  - Sapienza Università di Roma, Roma
- Kuwait University, Kuwait City, Kuwait
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador, Mexico City, Mexico
- Hospital Clínic Barcelona, Barcelona, Spain
- Sweden (2):
  - Linköping University, Linköping
  - Örebro University, Örebro
- Switzerland (2):
  - Clarunis Universitäres, Basel
  - Hôpitaux universitaires de Genève, Geneva
- United Kingdom (3):
  - Nuffield Health Bristol Hospital, Bristol
  - King's College Hospital, London
  - Queen Mary University, London

IPD SHARING:
Plan to Share IPD: Yes